CLINICAL TRIAL: NCT02149173
Title: Serial [F-18] Fluoroestradiol (FES) PET Imaging to Evaluate Endocrine-Targeted Therapy
Brief Title: F-18 FES PET/CT in Measuring Hormone Expression in Patients With Primary, Recurrent, or Metastatic Breast Cancer Undergoing Endocrine-Targeted Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to low accrual
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7184; NCI-2013-02342 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7184 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA042045 (NIH); U01CA148131 (NIH); RG1711032 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2014-05-01; First posted 2014-05-29 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Estrogen Receptor Positive; Recurrent Breast Carcinoma; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — 16-fluoroestradiol; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (F-18 FES PET/CT) (Experimental): Patients undergo F-18 FES PET/CT scan at baseline. Patients also undergo F-18 FES PET/CT and FDG PET/CT between 1-12 weeks after starting therapy, and then 1-12 weeks after the second FES PET/CT scan. Repeat FDG PET may be omitted in patients on selective estrogen receptor degrader.
  Interventions: Procedure: Computed Tomography; Drug: F-18 16 Alpha-Fluoroestradiol; Drug: Fludeoxyglucose F-18; Other: Laboratory Biomarker Analysis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo F-18 FES PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Procedure: Computed Tomography — Undergo FDG PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Drug: F-18 16 Alpha-Fluoroestradiol — Undergo F-18 FES PET/CT
  Other Names: 16 alpha-fluroestradiol-17 beta; F-18 FES; FES; Fluorine-18 16 alpha-fluoroestradiol; Fluoroestradiol F-18
Drug: Fludeoxyglucose F-18 — Undergo FDG PET/CT
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Positron Emission Tomography — Undergo F-18 FES PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Procedure: Positron Emission Tomography — Undergo FDG PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This clinical trial studies use of F-18 16 alpha-fluoroestradiol ([F-18] FES) positron emission tomography (PET)/computed tomography (CT) in measuring tumor hormone receptor expression in patients undergoing endocrine-targeted therapy for newly diagnosed breast cancer or breast cancer that has come back or spread to other places in the body. Comparing results of diagnostic procedures done before, during, and after hormone therapy may help measure a patient's response to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Measure the effect of endocrine targeted therapy on estrogen receptor (ER) expression and estradiol binding to the receptor using serial FES PET and fludeoxyglucose F-18 (FDG) PET.

SECONDARY OBJECTIVES:

I. Document the safety profile of FES PET in patients with breast cancer.

II. Examine associations between FES PET results and serial measurements of hormone or other levels in peripheral blood, as related to efficacy of endocrine-targeted therapy. Correlate FES PET uptake measures with histopathological assays and tumor microenvironment studies on biopsy specimens, if relevant to specific treatment regimen.

OUTLINE:

Patients undergo F-18 FES PET/CT scan at baseline. Patients also undergo F-18 FES PET/CT and FDG PET/CT between 1-12 weeks after starting therapy, and then 1-12 weeks after the second FES PET/CT scan. Repeat FDG PET may be omitted in patients on selective estrogen receptor degrader.

After completion of study, patients are followed up for up to 20 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult, non-pregnant patients with biopsy-proven or clinically obvious primary, recurrent or metastatic breast cancer
* Breast cancer from ER+ primary that is seen on other imaging tests; tumor ER expression must have been confirmed by immunohistocytochemistry of primary tumor or recurrent disease
* At least one site of disease 1.5 cm or greater is needed to meet the spatial resolution limits of PET imaging
* Patients must have been off tamoxifen or other estrogen receptor blocking agents for at least 6 weeks and off chemotherapy for 3 weeks for the initial baseline FES
* Patients must be selected for an endocrine targeted therapy regimen for treatment of their breast cancer by the referring oncologist; selected treatments may be part of experimental treatment protocols for which the patient would be separately consented
* Patients must be willing to undergo serial imaging procedures
* Patients must agree to allow access to clinical records regarding response to treatment and long term follow up

Exclusion Criteria:

* An inability to lie still for the tests
* Individuals weighing more than 300 lb; (this is the weight limit of the scanner table)
* Pregnant or lactating; women of childbearing potential with either a positive or no pregnancy test at baseline are excluded
* Any other life-threatening illness (e.g. serious, uncontrolled concurrent infection or clinically significant cardiac disease - congestive heart failure, symptomatic coronary artery disease, cardiac arrhythmia not well controlled with medication)
* Use of tamoxifen, Faslodex, diethylstilbestrol (DES) or any other ER blocking agent < 6 weeks or chemotherapy < 3 weeks prior to imaging scan
* Unwillingness or inability to give informed consent
* Uncontrolled diabetes mellitus (fasting glucose > 200 mg/dL)
* Adult patients who require monitored anesthesia for PET scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-09-15 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Linden, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (F-18 FES PET/CT)
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 23 patients were co-enrolled in a vorinostat therapy study. The remaining 6 patients were enrolled in studies involving potential estrogen receptor blocking therapy.
Arm/Group | Diagnostic (F-18 FES PET/CT)
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 12
Age, Continuous [Median (Full Range); unit: years] | 62 [32 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in F-18 16 Alpha-fluoroestradiol (FES) Standardized Uptake Value (SUV), Assessed by a One-sample Test of the Percent Change in FES SUV
Description: Uptake was quantified using lean body mass adjusted SUV (SULmean). The geometric mean was calculated for up to 3 lesions per patient. Systematic change in FES SULgmean between baseline and a second FES scan at approximately 2 or 8 weeks and a third FES scan was at approximately 8 weeks measured using a sign test where the median change is zero.
Time Frame: from time of first F-18 FES-PET/CT scan to time of second or third F-18 FES-PET/CT scan (approximately 2-8 weeks)
Population: 15/23 patients underwent a second FES PET/CT scan approximately 2 wks after starting potential ER modulating (vorinostat) therapy. 14/23 underwent a second or third FES PET/CT scan approximately 8 wks after starting vorinostat therapy. 6 patients underwent a second FES PET/CT scan between 2-8 wks after starting potential ER blocking therapy.
Measure: Median (Full Range); unit: percentage of change in SULgmean
Groups:
- FES-imaging After 2 Wks of ER Modulating (Vorinostat) Therapy: Patients undergo F-18 FES PET/CT and FDG PET/CT scans at baseline. Patients also undergo F-18 FES PET/CT between approximately 2 weeks after starting therapy
- FES-imaging After 8 Wks of ER Modulating (Vorinostat) Therapy: Patients undergo F-18 FES PET/CT and FDG PET/CT scans at baseline. Patients also undergo F-18 FES PET/CT between approximately 8 weeks after starting therapy
- FES-imaging After 2-8 Weeks of ER Blocking Therapy: Patients undergo F-18 FES PET/CT and FDG PET/CT scans at baseline. Patients also undergo F-18 FES PET/CT between approximately 2-8 weeks after starting estrogen receptor blocking therapy.
Arm/Group | FES-imaging After 2 Wks of ER Modulating (Vorinostat) Therapy | FES-imaging After 8 Wks of ER Modulating (Vorinostat) Therapy | FES-imaging After 2-8 Weeks of ER Blocking Therapy
Number analyzed (Participants) | 15 | 14 | 6
percentage of change in SULgmean | 8.7 [-22.2 to 54.7] | 1.9 [-61.5 to 113.9] | -60.3 [-91 to -14]

2. Primary Outcome: F-18 16 Alpha-fluoroestradiol (FES) Uptake
Description: Quantitative and qualitative measures of FES uptake for each disease site, a set of 1.5 cm diameter regions on three adjacent planes with the highest lesion FES uptake will be drawn to determine maximal FES uptake. Up to 10 sites seen on the static torso survey will be quantified. Lesions will qualitatively determined to be visible or not visible.
Time Frame: from time of first F-18 FES-PET/CT scan to time of second or third F-18 FES-PET/CT scan (approximately 2-8 weeks)
Population: quantitative and qualitative measure of FES positive lesions
Measure: Count of Units; unit: number of ER+ lesions
Units Other Than Participants: number of ER+ lesions
Groups:
- Quantitative Uptake: number of lesions with quantitative uptake (SULmax) above 0.85 (the value indicating a negative lesion)
- Qualitative Uptake: Number of lesions visually indicated as having FES uptake
Arm/Group | Quantitative Uptake | Qualitative Uptake
Number analyzed (Participants) | 29 | 29
Number analyzed (number of ER+ lesions) | 314 | 314
number of ER+ lesions | 281 | 243

3. Primary Outcome: Proportion of Patients Experienced a Threshold in Percentage Change, or Surpassed a Targeted Follow-up F-18 16 Alpha-fluoroestradiol (FES) Standardized Uptake Value (SUV)
Description: The number of patients showing a 20% increase in FES SULgmean compared to baseline at either 2 or 8 weeks using a 90% Wilson score binomial confidence interval.
Time Frame: from time of first F-18 FES-PET/CT scan to time of second or third F-18 FES-PET/CT scan (approximately 2-8 weeks)
Population: The patient arms different from Primary Outcome 1 because they are separated according to the type of therapy each group had (ER modulating or ER blocking), not by the number of FES scans that they had. Results are based on the change between 2 scans.
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Groups:
- FES With Potential ER Modulating Therapy (Vorinostat): Patients undergo F-18 FES PET/CT and FDG PET/CT scans at baseline. Patients also undergo F-18 FES PET/CT between 1-12 weeks after starting possible ER modulating therapy (vorinostat) and then 1-12 weeks after the second FES PET/CT scan.
- FES With Potential ER Blocking Therapy: Patients undergo F-18 FES PET/CT scan and FDG PET/CT at baseline. Patients also undergo F-18 FES PET/CT between 1-12 weeks after starting possible ER blocking therapy.
Arm/Group | FES With Potential ER Modulating Therapy (Vorinostat) | FES With Potential ER Blocking Therapy
Number analyzed (Participants) | 23 | 6
Proportion of participants | 0 [0 to 0.21] | 0 [0 to 0.31]

4. Secondary Outcome: Time to Disease Progression
Description: Months from the start of endocrine therapy to the time the patient is first recorded as having disease progression,
Time Frame: from start of therapy up to 20 years
Measure: Median (Full Range); unit: months
Arm/Group | FES With Potential ER Modulating Therapy (Vorinostat) | FES With Potential ER Blocking Therapy
Number analyzed (Participants) | 23 | 6
months | 2 [.1 to 21.2] | 5.6 [1.4 to 8.4]

ADVERSE EVENTS:
Time Frame: Patients were monitored after each injection of FES for 24 hours (up to 3 injections over approximately 8 weeks)
Description: This is an imaging study. No adverse events are expected or have been reported due to tracer injection or imaging. All deaths were due to the natural course of metastatic breast cancer after the time period that adverse events were collected for this study. Any adverse events due to therapy are reported in a separate study in which these patients were co-enrolled (ID: 7841) and Sanofi TED14856 (SAR439859)
Groups:
- Diagnostic (F-18 FES PET/CT): Patients undergo F-18 FES PET/CT scan at baseline. Patients also undergo F-18 FES PET/CT and FDG PET/CT between 1-12 weeks after starting therapy, and then 1-12 weeks after the second FES PET/CT scan.
Arm/Group | Diagnostic (F-18 FES PET/CT)
All-Cause Mortality (participants affected / at risk) | 24/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT02149173/Prot_SAP_000.pdf